CLINICAL TRIAL: NCT01552122
Title: A Phase III Randomized, Double-Blind, Active Comparator-Controlled Study to Evaluate the Effects of Odanacatib (MK-0822) on Bone Mineral Density, Tolerability, and Safety in the Treatment of Postmenopausal Women With Osteoporosis Previously Treated With Alendronate
Brief Title: Efficacy and Safety of Odanacatib in Postmenopausal Women Previously Treated With Alendronate (MK-0822-050)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-050
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis; Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — odanacatib; Alendronate; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Odanacatib (Experimental)
  Interventions: Drug: Odanacatib; Dietary Supplement: Cholecalciferol (Vitamin D3); Dietary Supplement: Calcium carbonate; Other: Placebo (alendronate)
- Alendronate (Active Comparator)
  Interventions: Drug: Alendronate; Other: Placebo (odanacatib); Dietary Supplement: Cholecalciferol (Vitamin D3); Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Drug: Odanacatib — Odanacatib 50 mg compressed tablet will be administered orally, once-a-week, for 24 months
  Other Names: MK-0822
  Arms: Odanacatib
Drug: Alendronate — Alendronate 70 mg compressed tablets will be administered orally, once-a-week, for 24 months; and a reduced dose of 35 mg will be administered in the same fashion to a subset of women, Japanese participants only, for the same 24-month duration.
  Other Names: Alendronate Sodium; Fosamax
  Arms: Alendronate
Other: Placebo (odanacatib) — One compressed tablet administered orally, once-a-week, for 24 months.
  Arms: Alendronate
Dietary Supplement: Cholecalciferol (Vitamin D3) — Two (2) 2800 IU compressed tablets administered orally, once-a-week, for 24 months.
Dietary Supplement: Calcium carbonate — Dietary and supplemental sources, taken as needed, to ensure a total daily calcium intake of approximately 1200 mg.
Other: Placebo (alendronate) — One compressed tablet administered orally, once-a-week, for 24 months.
  Arms: Odanacatib

SUMMARY:
This study will evaluate the therapeutic effects and safety of odanacatib on bone mineral density in osteoporotic postmenopausal women who were previously treated with alendronate.

ELIGIBILITY:
Inclusion Criteria:

* In good general health, and postmenopausal for at least 5 years or more
* Diagnosed with postmenopausal osteoporosis
* Currently taking alendronate for at least 3 years or more for the treatment of osteoporosis
* One hip free of orthopedic hardware (ie, total hip device, hip pin); anatomy is suitable to undergo a dual-emission X-ray absorptiometry (DXA) scan (ie, bone mineral density scan)
* Agrees to not to use any other medications for the treatment of osteoporosis except those provided to the participant during the study

Exclusion Criteria:

* Evidence of metabolic bone disorder
* History of malignancy (cancer) for 5 years or less
* Active thyroid disease that cannot be managed with medication
* Severe renal insufficiency (kidney disease), myocardial infarction, unstable angina, stroke or revascularization, untreated malabsorption syndrome, and/or osteonecrosis of the jaw, or anticipates undergoing a major dental procedure (e.g. dental extraction or implantation)
* Use, misuse, abuse, and/or addiction of illicit drugs and/or recent history

(within the last year) of drug or alcohol abuse or dependence

* Use of estrogen with or without progestin and/or raloxifene (ie, Evista®) or tamoxifen (ie, Nolvadex®, Tamofen®)
* Use of any oral bisphosphonate therapy other than alendronate; intravenous bisphosphonates (zoledronate, ibandronate, pamidronate); any form of calcitonin other than intranasal; anabolic steroids; and/or Strontium-containing products (ie, Osteovalin™)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Bone Mineral Density (BMD) of the Femoral Neck | Baseline and Month 24

SECONDARY OUTCOMES:
Percent Change from Baseline in BMD of the Lumbar Spine, Total Hip, and Trochanter | Baseline and Month 24